CLINICAL TRIAL: NCT05054777
Title: Chinese Multicenter Prospective Registry of Breast Cancer Patient Reported Outcome and Oncological Safety -Oncoplastic and Conventional BCS Cohort
Brief Title: Patient Report Outcome and Oncological Safety -Oncoplastic and Conventional BCS Cohort
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Zhiyong Yu, PhD, Shandong Cancer Hospital and Institute
Other Study IDs: ShandongCHI-18
Record Dates: First submitted 2021-09-14; First posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Patient Reported Outcome; Oncological Safety; Breast-conserving Surgery; Breast Cancer Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- oncoplastic breast-conserving surgery: The oncoplastic breast-conserving surgery were mainly those surgeries using volume displacement or volume replacement techniques
  Interventions: Procedure: oncoplastic breast-conserving surgery
- conventional breast-conserving surgery: The conventional breast-conserving surgery were performed without any oncoplastic operations
  Interventions: Procedure: conventional breast-conserving surgery

INTERVENTIONS:
Procedure: oncoplastic breast-conserving surgery — The patients received oncoplastic breast-conserving surgery, including volume displacement or volume replacement techniques
  Groups: oncoplastic breast-conserving surgery
Procedure: conventional breast-conserving surgery — conventional breast-conserving surgery without any oncoplastic operations
  Groups: conventional breast-conserving surgery

SUMMARY:
Breast-conserving surgery (BCS) is the traditional surgical treatment for early-stage breast cancer patients. There are evidences indicating that oncoplastic BCS could improve cosmetic outcomes and/or quality of life, and has similar oncological safety as conventional BCS does. However, these studies that focused on patient-reported outcomes and oncological safety were mainly from one institution or of small sample size. The variations across hospitals and regions were not fully analyzed. A multicenter prospective patient report outcome (PROs) and oncological safety will be planned to assess the PROs and safety for Chinese breast cancer patients who will undergo oncoplastic and conventional breast-conserving surgery (OBCS). This study follows the Helsinki Declaration and Chinese rules. All patients will be asked to sign the informed consent and will be followed up 24 months after operations. All data will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent signed;
2. Non-metastatic Breast cancer patients confirmed by pathology;
3. Adult (>18 years old, <80 years old);
4. Female;
5. Must undergo oncoplastic or conventional breast-conserving surgery;

Exclusion Criteria:

1. Inflammatory breast cancer, Stage IV breast cancer patients;
2. Have other malignant tumors;
3. Pregnancy women;
4. Have severe co-morbidities that compromise the patients' compliance to our protocol, or endanger the patients;
5. Refuse breast-conserving surgery.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — famale
Study Population: Non-metastatic breast cancer patients received surgical treatment in the hospital. The patients must fulfill indications of breast cancer surgery according to NCCN clinical guidelines, and do not have any absolute contraindications.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Patients' satisfaction：BREAST-Q score | Change from baseline at 6 months, 1 year and 2 years post-operatively
  The Breast-Q© is a patient reported outcome measure (PROM) for breast surgery that was rigorously developed to accurately measure patient reported satisfaction and quality of life (QOL). (http://www.mskcc.org/mskcc/shared/Breast-Q/index.html). The BREAST-Q was developed and validated with adherence to international guidelines. This PROM is composed of six scales that address: 1) psychosocial well-being, 2) physical well-being, 3) sexual well-being, 4) satisfaction with breasts, 5) satisfaction with outcome, and 6) satisfaction with care. Each module generates a Q-score on a 0-100 scale that can be used for quantitative analysis to enable statistical comparison of the pre- to the post-operative state.
EORTC QLQ-C30 | Change from baseline at 1 year and 2 years post-operatively
  The EORTC QLQ-C30 (Version 3) uses for the questions 1 to 28 a 4-point scale. The scale scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much"). Half points are not allowed. The range is 3. For the raw score, less points are considered to have a better outcome. The EORTC QLQ-C30 (Version 3) uses for the questions 29 and 30 a 7-points scale. The scale scores from 1 to 7: 1 ("very poor") to 7 ("excellent"). Half points are not allowed. The range is 6. First of all, raw score has to be calculated with mean values. Afterwards linear transformation is performed to be comparable. More points are considered to have a better outcome.
Health-related quality of life：EORTC QLQ-BR23 | Change from baseline at 1 year and 2 years post-operatively
  EORTC QLQ-BR-23 consists of 23 questions related to breast cancer. The questionnaire will be self-administered and will be given in patient's mother tongue. EORTC-QLQ-BR23: included functional scales (body image, sexual functioning, sexual enjoyment, and future perspective) and single item symptoms scales (systemic therapy side effects, breast symptoms, arm symptoms, and upset by hair loss). Questions used 4-point Likert scale (1 'Not at All' to 4 'Very Much'). Scores averaged and transformed to 0-100 scale. High score for functional scale=high/healthy level of functioning. High score for single item=high level of symptomatology/problems.
Recurrence-free survival | up to 24 months
  Recurrence-free survival (RFS) was calculated as time from breast cancer diagnosis until locoregional (LRRFS) or distant recurrence (DRFS) or death due to breast cancer, whichever came first

SECONDARY OUTCOMES:
Complication's ratio | up to 24 months
  Postoperative complications were classified following Clavien-Dindo Classification. Grade I complication (light inflammations, non-surgical haematoma or suffusion, seroma formation, partial skin/NAC loss, limited fat necrosis, SSI and lymphoedema) does not require medication or surgical treatment. Grade II complication is a Grade I complication that requires medication or surgical interaction (antibiotic therapy, resuture due SSI and multiple puncture due chronic seroma). Grade III complication requires invasive surgical action (haematoma evacuation, chronic inflammation which requires reoperation, severe fat necrosis, full skin/ NAC necrosis and wound dehiscense). Grade IV complication means temporary organ failure. Grade V complication is one that leads to death
Cosmetic results | Change from baseline at 1 year and 2 years post-operatively
  The primary aesthetic stage will be documented with standard photo documentation using valid BCCT. core software making it measurable which allows us to compare it. the photo documentation performed the standard way in 5 position (antero-posterior (ap), 45 degree oblique and 90 degree lateral), in ap direction both ways arms up and down with strict adherence to personal privacy policies. The mentioned software counts measurements regarding to the photo documentation and gives a 4-point rating scale (1: excellent, 2: good, 3: acceptable, 4: non-acceptable). These numerical results can be statistically analyzed. We use the Likert scale (1. definitely not, 2: no, 3: abstain, 4: agree, 4: definitely agree) for evaluating the subjective aesthetic outcome based on the photo documentation (preoperative, postoperative 4-6th weeks, 3rd months, every 6 months 5 years long). The results are collected and averaged.
Overall survival | up to 24 months
  Overall survival (OS) was defined as the time from beginning treatment to the time of death from any cause or the date of last contact if death was not recorded before the cutoff date.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Weber WP, Soysal SD, Fulco I, Barandun M, Babst D, Kalbermatten D, Schaefer DJ, Oertli D, Kappos EA, Haug M. Standardization of oncoplastic breast conserving surgery. Eur J Surg Oncol. 2017 Jul;43(7):1236-1243. doi: 10.1016/j.ejso.2017.01.006. Epub 2017 Jan 31. PMID 28214053